CLINICAL TRIAL: NCT01570764
Title: Intravenous Cyclophosphamide for the Treatment of Systemic Sclerosis Associated Interstitial Lung Disease
Brief Title: Cyclophosphamide Systemic Sclerosis Associated Interstitial Lung Disease
Acronym: SCLEROCYC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hôpital Claude-Huriez (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P081241; 2011-004709-26 (EudraCT Number)
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis; Scleroderma; Interstitial Lung Disease; Lung Fibrosis
Keywords: Systemic sclerosis; Interstitial lung disease; Worsening; Cyclophosphamide; Intravenous
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial; Pulmonary Fibrosis | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclophosphamide (Experimental): Prednisone 15 mg/d + monthly pulse cyclophosphamide 700 mg/m ² diminished to 600 mg/m ² in patients over 65 years or having a creatinine clearance lower than 30 ml/min for 12 months.
  Interventions: Drug: Cyclophosphamide
- Placebo (Placebo Comparator): Prednisone 15 mg/d + monthly pulse of placebo of cyclophosphamide. The posology and the methods of administration of the placebo of cyclophosphamide (NaCl) will be the same as those used for cyclophosphamide
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclophosphamide — Prednisone 15 mg/d + monthly pulse cyclophosphamide 700 mg/m ² diminished to 600 mg/m ² in patients over 65 years or having a creatinine clearance lower than 30 ml/min for 12 months.
  Arms: Cyclophosphamide
Drug: Placebo — Prednisone 15 mg/d + monthly pulse of placebo of cyclophosphamide. The posology and the methods of administration of the placebo of cyclophosphamide (NaCl) will be the same as those used for cyclophosphamide
  Arms: Placebo

SUMMARY:
By including in this study patients with significant worsening of their lung volumes and / or their DLCO (carbon monoxide diffusing capacity) in the previous year, on the basis of an open retrospective study we recently conducted, we hope to demonstrate that a strategy combining prednisone and intravenous cyclophosphamide therapy is accompanied by an increase in the frequency stabilization / improvement of lung volumes and / or DLCO of patients at 12 months of 15% in the placebo and prednisone cyclophosphamide 50% in cyclophosphamide and prednisone.We also hope to demonstrate significant decrease in the number of patients excluded for failure in the CYC arm as compared to the placebo arm.

DETAILED DESCRIPTION:
This is a randomized prospective multicenter study evaluating the efficacy against placebo of cyclophosphamide in combination with prednisone in the treatment of systemic sclerosis related interstitial lung disease. Patients will be allocated, after randomization into two groups receiving both corticosteroids: a group of patients receiving placebo of cyclophosphamide and a group of patients treated with cyclophosphamide. Cyclophosphamide will be administered IV at a dose of 0.7 g / m (maximum 1200 mg) every 4 weeks. In patients over 65 or if the creatinine clearance below 30 ml / min the dose should be reduced to 0.6 g / m². The duration of treatment with cyclophosphamide will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Signed informed consent
* Patient with systemic sclerosis fulfilling the ACR -American college of rheumatology - (Masi et al. 1980) and/or Leroy and Medsger (LeRoy and Medsger 2001) diagnostics criteria with worsening ILD (interstitial lung disease) identified on a high resolution chest CT scan and by worsening of forced vital capacity (FVC) and/or total lung capacity (TLC) ≥10% and/or worsening of DLCO ≥ 15% as compared to values obtained within the 3 to 18 months preceding inclusion (for DLCO, in the absence of pulmonary arterial hypertension upon echocardiography)
* Smokers may be included (DLCO must be performed at least 72h after stopping tobacco intake).
* Patients with pulmonary hypertension (mean pulmonary arterial pressure <35 mmHg upon right heart catheterisation) secondary to hypoxia due to pulmonary fibrosis will also be included into the study.
* Physical examination prior to inclusion into the study (results must be given to the patient).

  -: Contraception considered effective by the investigator (abstinence and / or oral contraception or mechanical) for women of childbearing age (negative pregnancy test at baseline)
* Affiliation with a mode of social security (profit or being entitled)

Exclusion Criteria:

* Prednisone prescribed a dose greater than 15 mg/d during the last 3 months.
* Scleroderma renal crisis or acute or critical limb ischemia within the last year preceding inclusion,
* Left ventricular ejection fraction below 40% evaluated by echocardiography.
* Out of proportion pulmonary hypertension (mean pulmonary artery pressure above 35 mmHg upon right heart catheterization).
* CYC treatment during the last 12 months.
* Allergy, hypersensitivity or documented adverse events or contra-indications to the drugs used in the study (cyclophosphamide, Uromitexan, corticosteroids, domperidone ...)
* Patients with a past history of cancer within four years before inclusion and/or a history of chemotherapy for cancer within four years before inclusion (in remission or without disease activity for more than four years). Inclusion is authorized for patients with a basal cell carcinoma in the last 5 years.
* Severe infection: sepsis, cellulitis, gangrene in the last three months
* Past history of cystitis related to cyclophosphamide treatment
* Association to another connective disease : systemic lupus erythematosus, syndrome of Gougerot-Sjögren with anti-SSA/SSB, mixed connective tissue disease
* Patient breastfeeding
* Failure to sign the informed consent or unable to consent
* Patient participating in another clinical trial
* Injection of Rituximab within 6 months preceding inclusion
* Methotrexate or Cellcept treatment at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | at 12 months
  Forced vital capacity at 12 months

SECONDARY OUTCOMES:
Mortality | at 12 months
Progression free survival | at 12 months
  Progression free survival
Carbon monoxide diffusing capacity (DLCO) | at 12 months
Treatment failure | at 12 months
  Failure of cyclophosphamide or placebo
Walk test distance | at 12 months
  Six minutes walk test distance, O2 desaturation and gradient between maximal and minimal SAO2 during the test
Dyspnea | at 12 months
  NYHA (Classification de la New York Heart Association), BDI (Beck Depression Inventory) and Borg index
Health Assessment Questionnaire | at 12 months
Quality of life | at 12 months
  Saint-Georges; SF-36
Chest CT (computed tomography) scan | at 12 months
  CT (computed tomography) scan abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mouthon, MD, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No